CLINICAL TRIAL: NCT02197260
Title: Antimicrobial Therapy as Adjunct to Periodontal Treatment: Effect of Timing on Clinical, Microbiological and Systemic Response
Brief Title: Antimicrobial Therapy as Adjunct to Periodontal Treatment: Effect of Timing
Acronym: GAR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Geneva, Switzerland (Other)
Responsible Party: Principal Investigator, Andrea Mombelli, Prof. Dr.med.dent., University of Geneva, Switzerland
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 320030-122089; 2008DR4228 (Other: Swissmedic)
Record Dates: First submitted 2014-07-18; First posted 2014-07-22 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Chronic Periodontitis
Keywords: Periodontitis; amoxicillin; metronidazole; case management
MeSH Terms: conditions — Chronic Periodontitis; Periodontitis | interventions — Metronidazole; Amoxicillin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Protocol A (Experimental): Antibiotics (3/d 500 mg metronidazole plus 375 mg amoxicillin for 7 days) during the first, non-surgical phase of periodontal therapy (T1), and placebo during the second, surgical phase (T2)
  Interventions: Drug: 3/d 500 mg metronidazole plus 375 mg amoxicillin for 7 days
- Protocol B (Active Comparator): Placebo during the first, non-surgical phase of periodontal therapy (T1), and antibiotics (3/d 500 mg metronidazole plus 375 mg amoxicillin for 7 days) during the second, surgical phase (T2)
  Interventions: Drug: 3/d 500 mg metronidazole plus 375 mg amoxicillin for 7 days

INTERVENTIONS:
Drug: 3/d 500 mg metronidazole plus 375 mg amoxicillin for 7 days — Systemic antibiotics after sub gingival mechanical debridement

SUMMARY:
It is common practice to carry out the therapy of periodontal diseases in two phases. In a first, non-surgical phase, bacterial deposits on tooth surfaces (plaque and calculus) are removed using a cleaning method called "scaling and root planing" (SRP). After three to six months the case is evaluated and, if necessary, further treatment is provided, usually taking a more aggressive, surgical approach. Beneficial effects of adjunctive systemic antibiotics on clinical outcomes have been shown repeatedly but specific indications for antibiotics in subgroups of diseased patients, and the optimal timing of antimicrobial therapy, continue to be issues of a long lasting controversy.This study assessed the differential outcomes of periodontal therapy supplemented with amoxicillin-metronidazole during either the non-surgical or the surgical treatment phase.

DETAILED DESCRIPTION:
Single center, randomized placebo controlled crossover clinical trial with a one-year follow-up. Eighty participants with Aggregatibacter actinomycetemcomitans-associated chronic or aggressive periodontitis were randomized into two treatment groups. A: Antibiotics (3/d 500 mg metronidazole plus 375 mg amoxicillin for 7 days) during the first, non-surgical phase of periodontal therapy (T1), and placebo during the second, surgical phase (T2). B: Placebo during T1, and antibiotics during T2. Persistence of sites with a probing depth (PD) >4 mm and bleeding on probing (BOP) was the primary outcome. Evaluations were made three months after T1, as well as 6 and 12 months after T2.

ELIGIBILITY:
Inclusion Criteria:

* Untreated moderate to advanced periodontitis (at least 4 teeth with a probing pocket depth (PD) >4 mm, clinical attachment loss of at least 2 mm and radiographic evidence of bone loss)
* Presence of at least 12 scorable teeth (not including 3rd molars, teeth with orthodontic appliances, bridges, crowns or implants)
* Aggregatibacter actinomycetemcomitans-positive

Exclusion Criteria:

* Systemic illnesses (i.e. diabetes mellitus, cancer, HIV, bone metabolic diseases or disorders that compromise wound healing, radiation or immunosuppressive therapy)
* Pregnancy or lactation
* Systemic antibiotics taken within the previous two months
* Use of non-steroid anti-inflammatory drugs
* Confirmed or suspected intolerance to 5-nitroimidazole-derivatives or amoxicillin subgingival SRP or surgical periodontal therapy in the last year

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Number of persisting pockets >4 mm bleeding upon probing | one year after therapy

SECONDARY OUTCOMES:
Pocket depth of sites with baseline PD >4 mm | one year

OTHER OUTCOMES:
Adverse events | one year

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Mombelli, Dr.med.dent., Principal Investigator — University of Geneva
Locations (1):
- University of Geneva School of Dental Medicine, Geneva, Canton of Geneva, Switzerland

REFERENCES:
- [Result] Almaghlouth AA, Cionca N, Cancela JA, Decaillet F, Courvoisier DS, Giannopoulou C, Mombelli A. Effect of periodontal treatment on peak serum levels of inflammatory markers. Clin Oral Investig. 2014 Dec;18(9):2113-21. doi: 10.1007/s00784-014-1187-4. Epub 2014 Jan 23. PMID 24452825
- [Derived] Giannopoulou C, Cionca N, Almaghlouth A, Cancela J, Courvoisier DS, Mombelli A. Systemic Biomarkers in 2-Phase Antibiotic Periodontal Treatment: A Randomized Clinical Trial. J Dent Res. 2016 Mar;95(3):349-55. doi: 10.1177/0022034515618949. Epub 2015 Nov 24. PMID 26604272